CLINICAL TRIAL: NCT02217852
Title: A Randomized, Open-label, Positive Drug Controlled Clinical Trials to Compare the Efficacy of Nitrendipine and Hydrochlorothiazide , Captopril Plus Hydrochlorothiazide and Beijing Hypotensive No.0 in Tibetan Hypertension
Brief Title: Treatment of Hypertension in Tibetan Adult Population
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xiaoping Chen, Deputy director of Department of Internal Medicine, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WestChinaH 20140701
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Hypertension
Keywords: hypertension; Tibetan; Nitrendipine; hydrochlorothiazide; captopril; Beijing hypotensive No.0
MeSH Terms: conditions — Hypertension | interventions — Nitrendipine; Hydrochlorothiazide; captopril, hydrochlorothiazide drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A1 nitrendipine (Experimental): this arm will include Tibetan patients with hypertension whose BP is higher than 140/90mmHg but lower than 160/100mmHg and nitrendipine will be added (dose range 10mg-20mg bid).
  Interventions: Drug: Nitrendipine
- A2 hydrochlorothiazide (Experimental): this arm will include Tibetan patients with hypertension whose BP is higher than 140/90mmHg but lower than 160/100mmHg and hydrochlorothiazide will be added (dose range 12.5mg-25mg)
  Interventions: Drug: Hydrochlorothiazide
- B1 captopril plus Hydrochlorothiazide (Experimental): this arm will include Tibetan patients with hypertension whose BP is higher than 160/100mmHg and captopril plus Hydrochlorothiazide will be added (dose range：captopril 25mg-50mg tid, Hydrochlorothiazide 12.5mg-25mg qd).
  Interventions: Drug: Captopril,Hydrochlorothiazide
- B2 Beijing hypotensive No.0 (Experimental): this arm will include Tibetan patients with hypertension whose BP is higher than 160/100mmHg and Beijing hypotensive will be added (dose range：Beijing hypotensive No.0 one pile qd or less ).
  Interventions: Drug: Beijing hypotensive No.0

INTERVENTIONS:
Drug: Nitrendipine — doses used range from 10-20mg po bid. Total duration would be until completion or study or medication intolerance.
  Arms: A1 nitrendipine
Drug: Hydrochlorothiazide — doses used range from 12.5-25mg po qd. Total duration would be until completion or study or medication intolerance.
  Arms: A2 hydrochlorothiazide
Drug: Captopril,Hydrochlorothiazide — doses used range from 25-50mg po tid for captopril and 12.5-25mg po qd for hydrochlorothiazide. Total duration would be until completion or study or medication intolerance.
  Arms: B1 captopril plus Hydrochlorothiazide
Drug: Beijing hypotensive No.0 — 1 pile po qd or less. Total duration would be until completion or study or medication intolerance.
  Other Names: compound hypotensive tablet
  Arms: B2 Beijing hypotensive No.0

SUMMARY:
Several surveys had revealed that Tibetan adults had high prevalence of hypertension. However, there was no research studying the antihypertensive effect of the known drugs in Tibetan. The main arms of our study were to determine if the efficacy of lowing blood pressure and protecting target organ damage differs between nitrendipine and Hydrochlorothiazide in mild hypertension in Tibetan, and to determine if the efficacy of lowing blood pressure and protecting target organ damage differs between captopril plus Hydrochlorothiazide and Beijing hypotensive No.0 in moderate and severe Tibetan hypertension.

DETAILED DESCRIPTION:
Several surveys had revealed that Tibetan adults had high blood pressure(BP)and prevalence of hypertension than other parts of China and were also higher than those in developed nations as well. For example, one study found that among Tibetan herdsmen 40 years and older, the prevalence of hypertension was 56% and the mean systolic blood pressure/diastolic blood pressure was 146.6/92.0mmHg. However, the rates of awareness, treatment, and control were dismally low.

The Tibetan have been living in the Tibetan Plateau. The special natural and social environment there，as well as ethnic ,may all be involved in the etiology of the high prevalence and effect the response to antihypertensive treatment. Nevertheless, few interventional studies have been done in Tibetan hypertensive patients. Therefore, the purpose of our study was to compare the blood pressure reduction between different antihypertensive drugs. Nitrendipine, hydrochlorothiazide, captopril and Beijing hypotensive No.0 (also named" compound hypotensive tablet") are selected, which are cheap and available in the Tibetan Plateau.

Nitrendipine, hydrochlorothiazide and captopril are the representatives of Dihydropyridines Calcium antagonists, diuretics, and angiotensin-converting enzyme inhibitors, respectively. They are all recommended as the first-line antihypertensive drug. Beijing hypotensive No.0 is produce by China Resources Double-crane Pharmaceutical company in China, and it is a fixed-dose combination containing reserpine 0.1mg, hydrochlorothiazide 12.5mg, dihydralazine sulfate 12.5mg, triamterene 12.5mg. Many studies conducted in China have demonstrated its efficacy and safety in lowing blood pressure.

After recruitment, participant will be grouped according to their BP. If BP<160/100mmHg, monotherapy is started. Patient is randomly assigned to receive nitrendipine 10mg bid or Hydrochlorothiazide 12.5mg qd. If BP≥160/100mmHg, Patient is randomly assigned to receive two drug combination therapy(captopril 25mg three times daily (tid) and Hydrochlorothiazide 12.5mg qd) or Beijing hypotensive No.0 one pile qd. During the following 12 months，each participant will take at least four visits at 1、3、6 and 12 months respectively. Goal BP for all participants was less than 140/90mmHg, achieved by titrating the assigned study drug and adding open-label agents when necessary. The maximum dosage is 20mg BID for nitrendipine, 25mg qd for Hydrochlorothiazide and 50mg tid for captopril. The dosage of Beijing hypotensive No.0 should not be added.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Tibetan, who have been living in the Tibetan Plateau since he/she was born.
2. Consistent with diagnosed hypertension, blood pressure, for 1-3 grade.
3. Aged 18-80 years old.
4. To sign informed consent.

Exclusion Criteria:

1. diagnosis of secondary hypertension
2. Hypertensive emergencies and urgencies
3. Malignant hypertension
4. Bilateral renal artery stenosis, Chronic Kidney Disease（CKD）, serum creatinine> 133μmol / L.
5. Suffering from congenital heart disease, rheumatic heart disease, hypertrophic cardiomyopathy, aortic stenosis.
6. Occurred within the past 6 months who had a stroke or transient ischemic attack (TIA), unstable angina, myocardial infarction, percutaneous transluminal coronary angioplasty (PTCA).
7. clinical significance of arrhythmia
8. Active liver disease, history of chronic persistent hepatitis, alanine aminotransferase（ALT）> upper limit of normal.
9. Pregnancy, pregnancy or breast-feeding women to prepare.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-01 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Change of Blood Pressure | 12 months
  Change of systolic blood pressure，diastolic blood pressure and mean arterial pressure from baseline to study end at 12 months.

SECONDARY OUTCOMES:
Change of target organ damage | 12 months
  Change of target organ damage(including estimated glomerular filtration rate, microalbuminuria, carotid intima-media thickness, arterial stiffness, left ventricular mass index) from baseline to study end at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Chen, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China